CLINICAL TRIAL: NCT06824844
Title: The Effect of Topical 0.05% Cyclosporine Eye Drops on Diabetic Patients with Dry Eye Disease
Brief Title: The Effect of 0.05% CsA Eye Drops on Diabetic Patients with Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CsA
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye
Keywords: dry eye; 0.05% cyclosporine; diabetes
MeSH Terms: conditions — Dry Eye Syndromes; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.05% cyclosporine eyedrops combined with artificial tear eyedrops (Experimental)
  Interventions: Drug: artificial tear eyedrops; Drug: 0.05% cyclosporine eyedrops
- artificial tear eyedrops (Active Comparator)
  Interventions: Drug: artificial tear eyedrops

INTERVENTIONS:
Drug: artificial tear eyedrops — The intervention group and control group were treated with artificial tear eyedrops four times a day.
Drug: 0.05% cyclosporine eyedrops — The intervention group was treated twice a day.
  Arms: 0.05% cyclosporine eyedrops combined with artificial tear eyedrops

SUMMARY:
The objective of this study is to observe the effects of 0.05% cyclosporine eye drops combined with artificial tears on patients with diabetes-associated dry eye, and to monitor changes in ocular surface characteristics and inflammatory cytokines in tears before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

I. Age: 50 to 70 years old; II. Gender: No restriction; III. Meets the diagnostic criteria for dry eye: Refer to the 2020 Chinese Expert Consensus on Diagnostic Criteria for Dry Eye.

IV. Meets the diagnostic criteria for diabetes: History of type 2 diabetes with a course of ≥5 years; Diagnosis refers to the 1999 WHO Diagnostic Criteria for Diabetes.

V. Provision of written informed consent.

Exclusion Criteria:

I. active ocular infection, ocular inflammation, active ocular allergy, severe blepharitis or obvious inflammation of the eyelid margin.

II. Uncontrolled systemic disease. III.Suffer from diseases that may affect corneal nerves, such as keratoconus, trigeminal neuralgia, allergic conjunctivitis, etc.

-

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
ocular surface disease index (OSDI) | from baseline to 3 months after treatment
  OSDI is one of the most frequently used questionnaires for evaluation of dry eye disease (DED). This includes 12 questions which measure the frequency of symptoms over the recent week, and the scores range from 0 to 100.
Tear break-up time (TBUT)(s) | from baseline to 3 months after treatment
  BUT is the time from normal blinking to the first appearance of a break in the tear film.
Corneal fluorescein staining (CFS) | from baseline to 3 months after treatment
  The degree of fluorescein staining of the cornea was evaluated using the National Eye Institute (NEI) scale of five corneal regions (central, superior, temporal, nasal, and inferior). The scores range from 0 to 15.
Schirmer I test (SIt) (mm/5 minutes) | from baseline to 3 months after treatment
  The Schirmer I test is performed using sterile strips without anesthesia. The strips are placed in the lateral part of the inferior fornix of the eye for 5min and the extent of tear flow down was measured in millimeters.
Lissamine green staining | from baseline to 3 months after treatment
  To grade the temporal zone, the subject looks nasally; to grade the nasal zone the subject looks temporally. The upper and lower conjunctiva can also be graded.

SECONDARY OUTCOMES:
corneal sensitivity (range, 60-0 mm) | from baseline to 3 months after treatment
  Corneal sensitivity will be measured in the right eye only using the Cochet-Bonnet aesthesiometer and the ascending method of limits to determine the threshold of stimulus detection.
the concentration of Interleukin-1β (IL-1β) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-1β levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-6 (IL-6) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-6 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-10 (IL-10) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-10 levels will be quantified by Luminex immunoassay.
the concentration of Interleukin-17A (IL-17A) (pg/ml) | from baseline to 3 months after treatment
  basal tears will be collected from the inferior meniscus of each subject to test this inflammatory cytokine. IL-17A levels will be quantified by Luminex immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No